CLINICAL TRIAL: NCT00156143
Title: GH Therapy in Partial GHD Adolescents : Evaluation of Efficacy Based on Body Composition and Comparison of 2 Different Doses of Genotonorm®. Open-Label, Randomised, Comparative, Controlled, Parallel-Group, Multi-Center Phase IIIB Clinical Trial.
Brief Title: Transition Study: Growth Hormone Therapy In Partial Growth Hormone Deficient Adolescents
Acronym: TAUBER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 307-MET-9002-016; A6281018
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2007-07-30 (Estimated); Status verified 2007-07

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Blood Specimen Collection; X-Rays

INTERVENTIONS:
Procedure: Blood sample
Procedure: Radiography

SUMMARY:
To evaluate in boys and girls the improvement in body composition under GH treatment in adolescents with CO-GHD who remain partially GHD after GH discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Males or females : Chronological age > or = 15 years and < or = 20 years for females
* Chronological age > or = 17 years and < or = 20 years for males
* GHD of childhood onset treated for at least 2 years
* Last GH injection at least 12 months before baseline visit

Exclusion Criteria:

* Turner's syndrome
* Chronic hepatic impairment as shown by GGT and / or ASAT and / or ALAT > 2 X ULN

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90
Dates: Start 2002-04; Study Completion 2005-04

PRIMARY OUTCOMES:
Change from baseline of the % of fat mass assessed by DEXA after 1 year of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer